CLINICAL TRIAL: NCT06077045
Title: Uptake of the Childhood Live Attenuated Influenza Vaccine (LAIV) and Influenza-related Healthcare Resource Use in England During the 2012 to 2022 Flu Seasons; a Retrospective, Observational Study in the CPRD and HES Databases
Acronym: INOCULATE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2560R00011
Record Dates: First submitted 2023-07-12; First posted 2023-10-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- LAIV Vaccinated cohort: All individuals receiving LAIV between 2 and <18 years within a given flu season between 2012 and 2020.
- Unvaccinated cohort: All individuals between 2 and <18 years with no record of influenza vaccinations in a given flu season

SUMMARY:
In 2013, the NHS started a vaccination program in some regions of England to provide free flu vaccines to children aged 2 years or older, and younger than 16 years. The program has since been rolled out across England. Most children are given a vaccine that is sprayed into their nose. In clinical trials, this vaccine has been shown to protect children from experiencing severe flu symptoms. It is important to describe how it is used, and what happens to children who receive it in the wider community. This evidence will help the NHS to check that the vaccine roll out runs as planned and produces the intended benefits.

This study aims to: (1) describe how many children each year receive flu vaccines, and describe the characteristics of children who are and aren't vaccinated for influenza; (2) test how often children receiving the vaccine see their GP or a hospital doctor for symptoms related to flu, compared to those who don't; and (3) to test what groups of children are more or less likely to receive a flu vaccine. To answer these objectives, the study will use the Clinical Practice Research Datalink, linked to Hospital Episode Statistics and the Office for National Statistics database.

DETAILED DESCRIPTION:
A Live Attenuated Influenza Vaccination (LAIV) has been offered to children through a rolling national program in England since 2013. Previous observational studies identified trends in LAIV uptake that varied with demographic and clinical profiles.

The general aim of this study is to provide up-to-date epidemiological evidence on the uptake of the influenza vaccines, and influenza related HCRU outcomes in children in England. The specific study objectives are given below.

Primary objective:

1. To evaluate the uptake of influenza vaccines in children aged ≥2 and <18 years in England between 2012 and 2020 for LAIV, QIV, and influenza vaccinations where the product is not specified

Secondary objectives:

2.1 To describe usage patterns of LAIV in England between 2012 and 2020. 2.2 To describe HCRU associated with laboratory confirmed influenza and/or influenza-like-illness (ILI) in England between 2012 and 2020 and assess the relative impact of LAIV on HCRU use of LAIV vs no vaccination 2.3 To describe demographics and clinical characteristics of individuals vaccinated with LAIV or not vaccinated against flu by any vaccine in each flu season between 2012 and 2020 2.4 To estimate a DAG aligned model for LAIV uptake in England based on demographic and clinical factors for each flu season and across multiple seasons between 2012 and 2020

The study will include all research eligible aged between ≥2 and <18 years in the study period, with 6 months of history in CPRD before their first influenza vaccination. It will use the Clinical Practice Research Datalink data (vaccinations, diagnoses, characteristics) linked to Hospital Episode Statistics (HCRU). Logistic regression analyses will be used to test for factors associated with vaccine uptake, and outcomes between vaccinated and unvaccinated children. The study will provide up-to-date epidemiological evidence on the uptake of LAIV and its impact on HCRU related to ILI in children in England. This may be used by the NHS for planning and evaluation of the childhood influenza vaccination program.

ELIGIBILITY:
The reference study cohort will include patients as follows:

* Aged ≥2 and <18 years at any time between 1 September 2012 and 30 April 2020
* Classified as eligible for inclusion in research analysis according to CPRD guidance

In each flu season, the following criteria apply:

Inclusion Criteria:

* Aged ≥6 months and <2 years on the 1st September
* Have a high-risk condition as listed in the Green Book.

Exclusion Criteria:

* Were deceased or had migrated out of their practice prior to the 1st September in the current influenza season.
* Were recorded has receiving both QIV and LAIV in the current influenza season.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will include all research eligible children born between the 1st January 1994 and 31st August 2020 (latest date at which a child can be aged 2 years or above in the study period and have at least six months follow up in the most recent data), with 6 months of medical history available in CPRD before their the 1st September in the first year they are aged 2 years or above. The childhood influenza programme has been conducted on a rolling basis since 2013. Classification of each child as eligible for the vaccine will therefore vary year on year depending on their age, GP practice location and presence of high-risk conditions.
Sampling Method: Non-Probability Sample
Enrollment: 12775880 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Uptake of influenza vaccination | Per flu season (defined as 1st September in a given year to the 30th April the following year )
  Proportion of eligible individuals receiving a flu vaccine (LAIV, QIV, other)

SECONDARY OUTCOMES:
GP consultations for ILI (influenza-like illness) | From vaccination date until the earliest of death, de-registration, or the end of the influenza season (30th April of the second calendar year the season spans).
  Rate of GP consultations for ILI per 100,000 person years.
Laboratory confirmed influenza | From vaccination date until the earliest of death, de-registration, or the end of the influenza season (30th April of the second calendar year the season spans).
  Rate of Laboratory confirmed influenza for ILI per 100,000 person years.
Admitted Patient Care (APC) episodes associated with ILI | From vaccination date until the earliest of death, de-registration, or the end of the influenza season (30th April of the second calendar year the season spans).
  Rate of Admitted Patient Care (APC) for ILI per 100,000 person years.
Accident and Emergency (A&E) attendances associated with ILI | From vaccination date until the earliest of death, de-registration, or the end of the influenza season (30th April of the second calendar year the season spans).
  Rate of A&E for ILI per 100,000 person years.
Outpatient attendances associated with ILI | From vaccination date until the earliest of death, de-registration, or the end of the influenza season (30th April of the second calendar year the season spans).
  Rate of Outpatient attendances associated with ILI per 100,000 person years.
Length of stay in APC for influenza and ILI | From vaccination date until the earliest of death, de-registration, or the end of the influenza season (30th April of the second calendar year the season spans).
  Average length of stay in hospital for influenza and ILI
Number of antibiotic prescriptions | From vaccination date until the earliest of death, de-registration, or the end of the influenza season (30th April of the second calendar year the season spans).
  Counts of antibiotic prescriptions
Number of antiviral prescriptions | From vaccination date until the earliest of death, de-registration, or the end of the influenza season (30th April of the second calendar year the season spans).
  Counts of antiviral prescriptions

CONTACTS AND LOCATIONS:
Locations (1):
- CPRD, London, United Kingdom

REFERENCES:
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2560R00011&attachmentIdentifier=e32fb856-d531-4d4a-a12b-2372fe020b6d&fileName=D2560R00011_redacted_CSR_Synopsis.pdf&versionIdentifier=